CLINICAL TRIAL: NCT04842461
Title: Presence of Psychopathy and Antisocial Personality Disorder as Well as Genetic Biomarkers and the Inhibition-prepulse Endophenotype in Elite Athletes
Brief Title: Mental Health, Addictions and Biomarkers in High Athletes Performance
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: Villarreal CF (Unknown)
Responsible Party: Principal Investigator, Isabel Almodóvar Fernández, PhD, Cardenal Herrera University
Other Study IDs: MHS
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mental Disorder; Anxiety; Depression; Substance Abuse; Pathological Gambling
Keywords: mental disorder; gambling; despression; anxiety
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Depression; Substance-Related Disorders; Gambling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sport is a privileged area to promote socialization and health values, such as companionship; a healthy lifestyle; cooperation to achieve common goals, and justice, rejecting unjustified advantages in competition. The concept of fair play is on which the development of those values pivots. From a holistic perspective, it is possible to define fair play, not only as a way to participate but also as a way of projecting people in life with values, assuming a set of behaviors that enhance a healthy and respectful sporting experience with opponents, the companions, the spectators, the referees and all the agents that take part in the sport practice.

DETAILED DESCRIPTION:
Sport is a privileged area to promote socialization and health values, such as companionship; a healthy lifestyle; cooperation to achieve common goals, and justice, rejecting unjustified advantages in competition. The concept of fair play is on which the development of those values pivots. From a holistic perspective, it is possible to define fair play, not only as a way to participate but also as a way of projecting people in life with values, assuming a set of behaviors that enhance a healthy and respectful sporting experience with opponents, the companions, the spectators, the referees and all the agents that take part in the sport practice.

Since 2018, joint actions have been carried out with the Villarreal de Fútbol Club, within the framework of the ENDAVANT agreement. Within these actions, it is proposed to develop different lines of research on sport and health. Within these lines, one of special relevance is that related to the risk of consumption of illicit substances and / or behavioral addictions, in elite athletes, since they are subjected to intense training days and stress situations derived from the demands of performance of professional competitive activity. On the other hand, recently published behavioral studies show that athletes who practice non-contact sports have a greater capacity to identify and assess emotions than athletes who practice contact sports and than those who practice contact sports show higher levels of physical aggression or verbal, and hostility or anger, than athletes who practice individual and non-contact sports.

ELIGIBILITY:
Inclusion Criteria:

* active athletes in the elite soccer competition from the Villarreal CF, who agree to be included in the study by signing an informed consent and who have a health profile made by the club's Medical Service.

Exclusion Criteria:

* athletes who are transferred to other clubs during the study period.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Elite football players from Spanish football league
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Common drugs | 2 years
  Describe the consumption of common drugs in elite athletes.
Identify other mental disorders | 2 years
  Identify other mental disorders differents than addictions and psychopathy in elite athletes.
Explore the consumption of new psychoactive substances | 2 years
  Explore the consumption of new psychoactive substances in elite athletes
Pathological gambling | 2 years
  Describe the study of behavioral addictions and video game addiction in elite athletes.
Mental disorders | 2 years
  Describe the presence of psychopathy and antisocial personality disorder
Genetic biomarkers | 2 years
  Describe genetic biomarkers endophenotype in elite athletes.
Dopping | 2 years
  Describe new dopping substances in elite atheletes.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Muñoz Macho, MD, Study Chair — Medical Services of Villarreal CF SAD
Locations (2):
- Spain (2):
  - Villarreal CF, Ciudad Real, Castellón
  - Villarreal CF, Villarreal, Castellón